CLINICAL TRIAL: NCT03086512
Title: A Randomized Prospective Pivotal Study Comparing Computerized Tomographic Progression of Bone Bridging After Subtalar Fusion Using Fully and Partially Threaded Screws
Brief Title: A Study Comparing Computerized Tomographic Progression of Bone Bridging After Subtalar Fusion Using Fully and Partially Threaded Screws
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Collaborators: Acumed, LLC (Industry)
Responsible Party: Principal Investigator, Alastair Younger, Orthopaedic Foot and ankle Surgeon, Professor, Head division of distal extremities, Department of Orthopaedics, University of British Columbia. Director of Foot and Ankle Research, St. Paul's Hospital., St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMD - 2015
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Subtalar Fusion

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups. Group I consists of 45 patients receiving a subtalar fusion with fully threaded screws (Acutrak 2® - 7.5). Group II consists of 45 patients receiving a subtalar fusion with partially threaded screws (Synthes® 7.3 Cannulated Screw).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group I (Active Comparator): Group I consists of 45 patients receiving a subtalar fusion with the Acutrak 2® - Fully Threaded Screw.
  Interventions: Device: Acutrak 2® - 7.5 Screw
- Group II (Sham Comparator): Group II consists of 45 patients receiving a subtalar fusion with the Partially Threaded Synthes® 7.3 Cannulated Screw.
  Interventions: Device: Synthes® 7.3 Cannulated Screw

INTERVENTIONS:
Device: Acutrak 2® - 7.5 Screw — The Acumed Acutrak 2® - 7.5 is a fully-threaded headless screw fixation, composed of 17 unique screw size options. The Acutrak 2® - 7.5 is available in sizes from 40 mm to 120 mm and is inserted using a 4.0 mm hex driver over a .094" guide wire. The Acutrak 2 Part Number is 30-0XXX and 30-0XXX-S.
  Arms: Group I
Device: Synthes® 7.3 Cannulated Screw — The Synthes® 7.3 mm Cannulated screws are available in three thread options: 16 mm, 32 mm or fully threaded. This study will use the partially threaded options. The screws can be placed by small diameter guide wires. They are composed of 316L stainless steel or titanium alloy (Ti-6Al-7Nb).
  Arms: Group II

SUMMARY:
The study was designed by the principal investigator, Dr. Alastair Younger, and the St. Paul's Hospital Foot and Ankle Research Group, who will conduct the study. The study is being funded by Acumed LLC, the manufacturer of the Health Canada approved Acutrak 2® - 7.5 fully threaded screw.

The purpose of this study is to assess and compare the effectiveness of fully threaded screws versus partially threaded screws in subtalar fusion, in order to determine the effect of the thread configuration on the success of the fusion procedure.

Efficacy will be assessed primarily by computed tomography (CT) analysis of percent bone bridging across the subtalar joint at both 12 and 24 weeks post-op. Outcome scores will also be administered to compare general health and foot function between the two groups at baseline and at multiple post-op follow-up visits. Additional resource utilization (i.e. additional clinic and/or hospital admissions) will also be compared between the two groups post-op.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 19 years of age.
* The subject is considered to be skeletally mature.
* The subject qualifies for subtalar fusion based on physical examination and/ or past medical history including isolated osteoarthritis, post-traumatic, degenerative, or rheumatoid arthritis of the ankle.
* The subject experiences severe pain in the subtalar joint that could not be cured with non-operative treatment options.
* The patient may undergo a subtalar fusion as part of a triple arthrodesis.
* The patient has a normally functioning ankle joint, a solidly fused ankle joint, or a well-functioning ankle joint replacement.
* The patient may have forefoot pathology addressed by either prior or concurrent surgery (osteotomies or fusions).
* An ankle joint replacement or ankle joint fusion may be performed during the same sitting.
* The patient consented for either an arthroscopic or open procedure.
* The subject is able to comply with all post-operative evaluations and visits.
* The subject consents to and will receive either a cancellous autograft bone graft or synthetic bone graft substitute

Exclusion Criteria:

* The subject has:

  1. Severe osteoporosis
  2. Neuromuscular impairment
  3. Prior infection in the affected joint
* The subject currently has acute infections that, in the opinion of the Investigator, may complicate healing.
* The subject has a known sensitivity or allergic reaction to the screw material.
* The subject has insufficient bone stock or bone quality to support the screws.
* The subject has a major risk factor for non-union (ex. poorly controlled diabetes or current smoker).
* The subject is undergoing a revision of a prior subtalar fusion.
* The subject has a BMI of > 50 kg/m2.
* The subject is known to be pregnant, or plans to become pregnant during the study period
* The investigator judges the subject to be unable or unlikely to remain compliant to follow-up due to a physical or mental condition (ex. currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.).
* The subject is unable to provide informed consent.
* The subject is unable to communicate with the research team.
* The subject is unable to comply with follow-up.
* The subject has a history of substance addiction (e.g. recreational drugs, narcotics, or alcohol) within 12 months prior to screening for study entry
* The subject is a prisoner, or is known or suspected to be transient
* The subject either does not consent to or will not be receiving either a cancellous autograft bone graft or synthetic bone graft substitute
* The subject will be receiving a structural autograft or allograft (such as a femoral head graft or tri cortical iliac crest graft) to fill a defect greater than 1cm3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-04-21 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative CT Scans: 12 Week Width of Joint | Measurements will be assessed at 12 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * For each observer at the time-point, each slice of the CT scan will be reviewed and the width of the joint will be measured.
Post-operative CT Scans: 12 Week Width of Bone Bridging | Measurements will be assessed at 12 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * For each observer at the time-point, each slice of the CT scan will be reviewed and the width of bone bridging will be measured.
Post-operative CT Scans: 12 Week Width of Any Fixation Hardware | Measurements will be assessed at 12 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * For each observer at the time-point, each slice of the CT scan will be reviewed and the width of any fixation hardware will be measured.
Post-operative CT Scans: 24 Week Width of Joint | Measurements will be assessed at 24 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * For each observer at the time-point, each slice of the CT scan will be reviewed and the width of the joint will be measured.
Post-operative CT Scans: 24 Week Width of Bone Bridging | Measurements will be assessed at 24 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * For each observer at the time-point, each slice of the CT scan will be reviewed and the width of bone bridging will be measured.
Post-operative CT Scans: 24 Week Width of Any Fixation Hardware | Measurements will be assessed at 24 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * For each observer at the time-point, each slice of the CT scan will be reviewed and the width of any fixation hardware will be measured.
Post-operative CT Scans: 12 Week Bone Bridging | Measurements will be assessed at 12 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * The percent of bone bridging will be calculated for each slice.
Post-operative CT Scans: 24 Week Bone Bridging | Measurements will be assessed at 24 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * The percent of bone bridging will be calculated for each slice.
Post-operative CT Scans: 12 Week Group Average Comparisons | Measurements will be assessed at 12 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * The averages of all coronal slices for the three observers (6 readings per 12 week post-operative CT scan) will be compared between the two study groups.
Post-operative CT Scans: 24 Week Group Average Comparisons | Measurements will be assessed at 24 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * The averages of all coronal slices for the three observers (6 readings per 24 week post-operative CT scan) will be compared between the two study groups.
Post-operative CT Scans: 12 Week Inter- and Intra Observer Reliability | Measurements will be assessed at 12 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * The averages of all slices in the coronal plane will be compared between the three observers at 12 weeks to determine the inter- and intra- observer reliability of the measurements.
Post-operative CT Scans: 24 Week Inter- and Intra Observer Reliability | Measurements will be assessed at 24 weeks post-operation.
  This outcome measure is to compare bone bridging between full thread versus partial thread screw.
  * The coronal images will have the area of the screw masked and will be reviewed by three independent, trained, and blinded observers.
  * The averages of all slices in the coronal plane will be compared between the three observers at 24 weeks to determine the inter- and intra- observer reliability of the measurements.

SECONDARY OUTCOMES:
Ankle Osteoarthritis Scale (AOS) | Outcome will be administered 5 times per patient: within 30 days of surgery, 6 weeks post-op, 12 weeks post-op, 24 weeks post-op and 52 weeks post-op.
  This questionnaire assesses pain and difficulty in both the left and right ankle.
Musculoskeletal Outcomes Data Evaluation and Management System (MODEMS) including Short Form 36 Health Survey (SF-36) | Outcome will be administered 5 times per patient: within 30 days of surgery, 6 weeks post-op, 12 weeks post-op, 24 weeks post-op and 52 weeks post-op.
  This questionnaire assesses multiple aspects patient health such as comorbidities, expectations/satisfaction, physical component score and mental component score. These measures and scores are values on a unitless scale.
Foot and Ankle Ability Measure (FAAM) | Outcome will be administered 5 times per patient: within 30 days of surgery, 6 weeks post-op, 12 weeks post-op, 24 weeks post-op and 52 weeks post-op.
  This questionnaire assesses activities of daily living and sports subscales.
Radiographic assessments performed pre-operatively and post-operatively | There are 4 assessments time points: within 30 days of surgery, 6 weeks post-op, 12 weeks post-op, and 52 weeks post-op.
  X-rays will be completed to confirm the status of the implanted study device. The x-rays will be assessed for component location and subsidence of the implanted screws and other radiographic parameters including radiolucencies, osteolysis, and hypertrophy.
Resource utilization between the groups including extra clinic visits, any reoperations within the study period, and any additional days in hospital during the study period | Outcome will be measured through study completion, an average of 1 year post-operation per patient.
  Additional clinic visits, post-operative hospital admissions, and re-operations will be recorded as part of assessment of health services and resource utilization. The total number additional resources will be recorded.
Relationship between disease specific outcome scores (AOS and FAAM) and degree of bone bridging | Outcome will be measured after AOS/FAAM outcome scores and degree of bone bridging is assessed for each patient, at approximately 1 year post-operation. .
  The relationship between questionnaire outcome scores and degree of bone bridging will be assessed. Questionnaire outcome scores are values on a unitless scale, while bone bridging is a percentage. The relationship is a single unit measure derived from the relationship between the outcome value and bone bridging percentage.
Inter and intra observer reliability of the percent bone healing measured on sagittal and coronal views | Measurements will be assessed at same time points as CT scans, at 12 and 24 weeks post-operation.
  The CT scan measurements will be assessed for reliability. Averages of all slices in the coronal and sagittal plane will be compared between the three observers on two occasions to determine the inter- and intra- observer reliability of the measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada